CLINICAL TRIAL: NCT00000522
Title: Treatment of Mild Hypertension Study (TOMHS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 41; R01HL034767 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension; Vascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension; Vascular Diseases | interventions — Diet, Sodium-Restricted; Diet, Reducing; Exercise; Ethanol; Chlorthalidone; Acebutolol; Doxazosin; Amlodipine; Enalapril

INTERVENTIONS:
Behavioral: diet, sodium-restricted
Behavioral: diet, reducing
Behavioral: exercise
Behavioral: alcohol restriction
Drug: chlorthalidone
Drug: acebutolol
Drug: doxazosin
Drug: amlodipine
Drug: enalapril

SUMMARY:
To compare the effects of nonpharmacologic therapy alone with those of one of five active drug regimens combined with non-pharmacologic therapy, for long- term management of patients with mild hypertension.

DETAILED DESCRIPTION:
BACKGROUND:

Dietary sodium reduction has a mild effect on the reduction of hypertension. Weight loss, while achievable in the short-run with diet alone, may also have only mild effects on hypertension and is very difficult to maintain with diet and/or behavior modification. Alteration of patients' lifestyles to decrease excessive alcohol intake is somewhat controversial. Medications, on the other hand, have clear benefits in terms of blood pressure lowering, and in the case of diuretics and beta-blockers, reduction in cardiovascular morbidity and mortality. However, there is concern about their justified use in mild hypertension since each one has side effects, some of which may have long-term implications, such as alteration in serum lipids. Newer classes of drugs--calcium antagonists, angiotensin converting enzyme inhibitors, alpha blockers--had not previously been compared long-term with diuretics and beta-blockers.

DESIGN NARRATIVE:

TOMHS I enrolled 902 men and women to determine the feasibility of a larger trial. Participants were randomized in a double-blind manner to one of six treatment groups and within two strata. Stratum I was for participants not on antihypertensive drugs and Stratum II for those on antihypertensive drugs at initial screening. There were six treatment arms: placebo, a diuretic (chlorthalidone), a beta-adrenergic blocking agent (acebutolol), an alpha blocker (doxazosin mesylate), a calcium antagonist (amlodipine maleate), and an angiotensin converting enzyme inhibitor (enalapril maleate). All participants received a lifestyle intervention program that included reduction of sodium chloride and alcohol intake as well as weight reduction and increase in physical activity. All participants were followed for at least 48 months, with an average of 54 months. The primary endpoint was lowering of blood pressure. The treatments were also compared for effects on blood chemistries including lipoproteins, echocardiographic left ventricular mass, ventricular ectopic activity and ST-T changes of ischemia as measured by ambulatory ECG monitoring, side effects, and quality of life. Randomization took place between October 1986 and March 1988. Active follow-up ended in March-April 1992. Data analysis ended in May 1994.

ELIGIBILITY:
Men and women, ages 45 to 69, with mild hypertension (diastolic blood pressure of 90-99 mm Hg at two of three visits for untreated individuals. Patients who received drug therapy must have had a DBP less than 95 mm Hg two to four weeks after drug.

Ages: 45 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1985-08; Study Completion 1994-05

CONTACTS AND LOCATIONS:
Overall Officials: Richard Grimm — University of Minnesota

REFERENCES:
- [Background] Mascioli SR, Grimm RH Jr, Neaton JD, Stamler J, Prineas RJ, Cutler JA, Elmer PJ, McDonald R, Schnaper H, Schoenberger J. Characteristics of participants at baseline in the Treatment of Mild Hypertension Study (TOMHS). Am J Cardiol. 1990 Sep 25;66(9):32C-35C. doi: 10.1016/0002-9149(90)90760-x. PMID 2220647
- [Background] The treatment of mild hypertension study. A randomized, placebo-controlled trial of a nutritional-hygienic regimen along with various drug monotherapies. The Treatment of Mild Hypertension Research Group. Arch Intern Med. 1991 Jul;151(7):1413-23. doi: 10.1001/archinte.151.7.1413. PMID 2064494
- [Background] Liebson PR, Grandits G, Prineas R, Dianzumba S, Flack JM, Cutler JA, Grimm R, Stamler J. Echocardiographic correlates of left ventricular structure among 844 mildly hypertensive men and women in the Treatment of Mild Hypertension Study (TOMHS). Circulation. 1993 Feb;87(2):476-86. doi: 10.1161/01.cir.87.2.476. PMID 8425295
- [Background] Neaton JD, Grimm RH Jr, Prineas RJ, Stamler J, Grandits GA, Elmer PJ, Cutler JA, Flack JM, Schoenberger JA, McDonald R, et al. Treatment of Mild Hypertension Study. Final results. Treatment of Mild Hypertension Study Research Group. JAMA. 1993 Aug 11;270(6):713-24. PMID 8336373
- [Background] Black HR. Treatment of mild hypertension. The more things change.. JAMA. 1993 Aug 11;270(6):757-9. No abstract available. PMID 8336380
- [Background] Flack JM, Neaton JD, Daniels B, Esunge P. Ethnicity and renal disease: lessons from the Multiple Risk Factor Intervention Trial and the Treatment of Mild Hypertension Study. Am J Kidney Dis. 1993 Apr;21(4 Suppl 1):31-40. doi: 10.1016/s0272-6386(12)80859-6. PMID 8465834
- [Background] Elmer PJ, Grimm R Jr, Laing B, Grandits G, Svendsen K, Van Heel N, Betz E, Raines J, Link M, Stamler J, et al. Lifestyle intervention: results of the Treatment of Mild Hypertension Study (TOMHS). Prev Med. 1995 Jul;24(4):378-88. doi: 10.1006/pmed.1995.1062. PMID 7479629
- [Background] Stamler J, Prineas RJ, Neaton JD, Grimm RH, McDonald RH, Schnaper HW, Schoenberger JA, Elmer PJ, Cutler JA. Background and design of the new U.S. trial on diet and drug treatment of "mild" hypertension (TOMHS). Am J Cardiol. 1987 May 29;59(14):51G-60G. doi: 10.1016/0002-9149(87)90158-5. PMID 3296721
- [Background] Prineas RJ, Grimm R, Grandits G, et al: The Effect of Dietary Sodium and Body Weight on Echocardiographic Measures of Left Ventricular Mass Among Treated Hypertensive Men and Women: Four-Year Change in the TOMHS Study. Nieren-und Hochdruck-krankheiten, Jahrgang 23:S14-S21, 1994.
- [Background] Grandits GA, Liebson PR, Dianzumba S, Prineas RJ. Echocardiography in multicenter clinical trials: experience from the Treatment of Mild Hypertension Study. Control Clin Trials. 1994 Oct;15(5):395-410. doi: 10.1016/0197-2456(94)90035-3. PMID 8001359
- [Background] Liebson PR, Grandits GA, Dianzumba S, Prineas RJ, Grimm RH Jr, Neaton JD, Stamler J. Comparison of five antihypertensive monotherapies and placebo for change in left ventricular mass in patients receiving nutritional-hygienic therapy in the Treatment of Mild Hypertension Study (TOMHS). Circulation. 1995 Feb 1;91(3):698-706. doi: 10.1161/01.cir.91.3.698. PMID 7828296
- [Background] Crow RS, Prineas RJ, Rautaharju P, Hannan P, Liebson PR. Relation between electrocardiography and echocardiography for left ventricular mass in mild systemic hypertension (results from Treatment of Mild Hypertension Study). Am J Cardiol. 1995 Jun 15;75(17):1233-8. PMID 7778546
- [Background] Grimm RH Jr, Flack JM, Grandits GA, Elmer PJ, Neaton JD, Cutler JA, Lewis C, McDonald R, Schoenberger J, Stamler J. Long-term effects on plasma lipids of diet and drugs to treat hypertension. Treatment of Mild Hypertension Study (TOMHS) Research Group. JAMA. 1996 May 22-29;275(20):1549-56. doi: 10.1001/jama.1996.03530440029033. PMID 8622245
- [Background] Grimm RH Jr, Grandits GA, Prineas RJ, McDonald RH, Lewis CE, Flack JM, Yunis C, Svendsen K, Liebson PR, Elmer PJ. Long-term effects on sexual function of five antihypertensive drugs and nutritional hygienic treatment in hypertensive men and women. Treatment of Mild Hypertension Study (TOMHS). Hypertension. 1997 Jan;29(1 Pt 1):8-14. doi: 10.1161/01.hyp.29.1.8. PMID 9039073
- [Background] Lewis CE, Grandits A, Flack J, McDonald R, Elmer PJ. Efficacy and tolerance of antihypertensive treatment in men and women with stage 1 diastolic hypertension. Results of the Treatment of Mild Hypertension Study. Arch Intern Med. 1996 Feb 26;156(4):377-85. PMID 8607723
- [Background] Grimm RH Jr, Grandits GA, Cutler JA, Stewart AL, McDonald RH, Svendsen K, Prineas RJ, Liebson PR. Relationships of quality-of-life measures to long-term lifestyle and drug treatment in the Treatment of Mild Hypertension Study. Arch Intern Med. 1997 Mar 24;157(6):638-48. PMID 9080918
- [Background] Ganguli MC, Grimm RH Jr, Svendsen KH, Flack JM, Grandits GA, Elmer PJ. Urinary sodium and potassium profile of blacks and whites in relation to education in two different geographic urban areas. TOMHS Research Group. Treatment of Mild Hypertension Study. Am J Hypertens. 1999 Jan;12(1 Pt 1):69-72. doi: 10.1016/s0895-7061(98)00218-0. PMID 10075387
- [Background] Ganguli MC, Grimm RH Jr, Svendsen KH, Flack JM, Grandits GA, Elmer PJ. Higher education and income are related to a better Na:K ratio in blacks: baseline results of the Treatment of Mild Hypertension Study (TOMHS) data. Am J Hypertens. 1997 Sep;10(9 Pt 1):979-84. doi: 10.1016/s0895-7061(97)00162-3. PMID 9324102
- [Background] Grandits GA, Grimm RH Jr, Prineas RJ, Grambsch P, Holland LA. Obtaining event status at the close of the Treatment of Mild Hypertension Study: methods and implication for other trials. Control Clin Trials. 2001 Feb;22(1):56-61. doi: 10.1016/s0197-2456(00)00121-5. PMID 11165424